CLINICAL TRIAL: NCT01096602
Title: Blockade of PD-1 in Conjunction With the Dendritic Cell/AML Vaccine Following Chemotherapy Induced Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Medivation, Inc. (Industry); The Leukemia and Lymphoma Society (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-412
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Myelogenous Leukemia; AML
Keywords: Dendritic Cell/AML vaccine; CT-011
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): DC AML Fusion Vaccine
  Interventions: Biological: DC AML Vaccine

INTERVENTIONS:
Biological: DC AML Vaccine — Group 1: 2-3 doses of the vaccine at 4 week intervals

SUMMARY:
Acute myelogenous leukemia (AML) arises from leukemia stem cells that are difficult to eradicate and serve as a reservoir for disease relapse following chemotherapy. A promising area of investigation is the development of immunotherapeutic approaches that stimulate the immune system to recognize leukemia stem cells as foreign and eliminate them. The purpose of this research study is to determine the safety of the Dendritic Cell AML Fusion Vaccine (DC AML vaccine) after participants have achieved a remission with chemotherapy. In this clinical trial, patients are treated with a tumor vaccine alone following standard of care chemotherapy. The DC AML vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells. It is hoped that DC AML vaccine will prevent or delay the disease from coming back.

DETAILED DESCRIPTION:
* On this study participants will receive the DC AML vaccine and GM-CSF 4-8 weeks after completion of chemotherapy for acute myelogenous leukemia (AML). GM-CSF is a drug that stimulates white blood cells and is given with the DC AML Vaccine in an effort to enhance the effect of the vaccine. Participants will receive 2-3 doses of the vaccine at 4 week intervals.
* All participants will undergo the following procedures: Isolation of tumor cells by either bone marrow biopsy or blood draw; Initial chemotherapy for AML with standard therapy; Leukopheresis (collection of white blood cells from the blood).
* All participants will also have blood tests, a physical exam, and an electrocardiogram prior to each dose of vaccine.
* Four weeks following the final vaccination, participants will undergo a skin test called "delayed-type hypersensitivity" (DTH). This is an injection of the tumor cells under the skin to measure how the immune system responds. The tumor cells are broken up and irradiated to prevent their growth.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* Patients with AML at initial diagnosis or at first relapse
* 18 years of age or older
* ECOG Performance Status 0-2
* Life expectancy of greater than 9 weeks
* Laboratory values within limits outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Prior to Cell Collections for Dendritic Cell Generation:

* Patients must have obtained complete remission with chemotherapy defined by the absence of circulating blasts, and less then 5% blasts on bone marrow examination following hematopoietic recovery
* Resolution of all chemotherapy related Grade III-IV toxicity as per CTC criteria 4.0
* Laboratory values as outlined in the protocol
* For patients with evidence of minimal residual disease prior to vaccination, assessment of minimal residual disease status by cytogenetics or FISH will be followed post vaccination

Prior to Post-Chemotherapy Immunotherapy:

* Resolution of all chemotherapy related grade III-IV toxicity
* Laboratory values as outlined in the protocol
* At least 2 doses of fusion vaccine produced

Exclusion Criteria:

Screening:

* Active or history of autoimmune disorders/conditions including Type 1 diabetes. Type II diabetes, vitiligo or stable hyperthyroidism will not be considered exclusion criteria
* HIV positive
* Significant cardiac disease characterized by symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia
* Pregnant women
* Individuals with a history of a different malignancy are ineligible except for circumstances outlined in the protocol document

Prior to Cell Collection for Dendritic Cell Generation:

* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Patients who choose to proceed with allogeneic or autologous transplant at the time of remission will not be vaccinated and will come off study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2023-12 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Toxicity | 2 years
  To assess the toxicity associated with treating AML patients with DC/AML fusion cells in the post-chemotherapy setting

SECONDARY OUTCOMES:
Immune Response | 2 years
  To explore immunological response to DC/AML fusion vaccination in patients who have achieved a chemotherapy-induced remission.
T-cell and Immune Response | 2 years
  To correlate levels of circulating activated and regulatory T cells with immunologic response
Disease Response | 2 years
  To define anti-tumor effects by determining time to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722